CLINICAL TRIAL: NCT04590690
Title: Gut Microbiome and Sex as Risk Factors for Kidney Stones After Bariatric Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB19-1534
Record Dates: First submitted 2020-09-25; First posted 2020-10-19 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Bariatric Surgery Candidate
Keywords: bariatric surgery; kidney stones
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roux-en-y gastric bypass subjects (Experimental): Inclusion Criteria: Age 18-70. Participants pre-Roux-en-y gastric bypass (RYGB) who are approved and planned for Roux-en-y gastric bypass surgery in the Bariatric Surgery Center at the UCM.
  Exclusion Criteria: Patients with primary kidney diseases, kidney stone disease, or kidney impairment (eGFR < 90). Patients with known bladder voiding problems.
  Participants will complete a diet record and a 24-hour urine collection both before and after surgery.
  Participants will consume a 3 day fixed diet and present to the clinical research center for timed blood and urine draws. They will do this before and twice after (1 month and 1 year) surgery.
  Interventions: Other: Special diet
- Sleeve gastrectomy subjects (Experimental): Inclusion Criteria: Age 18-70. Participants pre-sleeve gastrectomy who are approved and sleeve gastrectomy in the Bariatric Surgery Center at the UCM.
  Exclusion Criteria: Patients with primary kidney diseases, kidney stone disease, or kidney impairment (eGFR < 90). Patients with known bladder voiding problems.
  Participants will complete a diet record and a 24-hour urine collection both before and after surgery.
  Participants will consume a 3 day fixed diet and present to the clinical research center for timed blood and urine draws. They will do this before and twice after (1 month and 1 year) surgery.
  Interventions: Other: Special diet

INTERVENTIONS:
Other: Special diet — The research clinic will provide subjects with a special diet for six days. After six days of isocaloric sodium, calcium and fluid intake, the study team will analyze three sequential 24-hour urine compositions including supersaturation of calcium oxalate, calcium, and urine volume, as well as stool collections. We will also evaluate components of 24-hour urine composition, specifically supersaturation, and the microbial contributions to urinary composition in 72-hour stool samples simultaneously collected using shot-gun metagenomic sequencing in men and women 1 year after surgery.

SUMMARY:
This is a single-center study that aims to better understand how diet and sex affect the risk of kidney stones in people who have had gastric bypass surgery. Subjects will be asked to follow a special (clinic-provided) diet for six days and come to a research clinic for 3 study visits.

DETAILED DESCRIPTION:
Experimental Design: We will determine sex differences in 24-hour urine supersaturation (SS) with respect to calcium oxalate (CaOx) in Roux-en-Y Gastric Bypass (RYGB) and sleeve gastrectomy patients and the correlation of microbial species and their metabolic pathways with urine oxalate. This will be determined under the conditions of an isocaloric, standardized sodium (200 mmol/day), calcium, potassium, macronutrient distribution. We will recruit subjects from the Bariatric Surgery Clinic at The University of Chicago Medical Center.

Location: The study will take place at participants' homes (Periods 1, 4) and in the University of Chicago Medicine (UCM) Clinical Research Center. (Periods 2, 3, 5).

Study period:

The study will consist of 5 separate periods. Periods 1 and 2 will be before surgery and periods 3-5 will occur after surgery. Periods 1 and 4 will last three days and periods 2, 3, and 5 will last four days, three of which are at home and a fourth (half-day) in the Clinical Research Center (CRC).

Study period 1 will occur prior to RYGB or specific gravity (SG) in the participant's home. Each participant will provide a three-day diet record and complete a 1.5-hour phone call with the CRC dietician and one 24-hour urine collection (on day three). Urine collection kits will be couriered directly to home and couriered back to the Kidney Stone Lab after completion.

Study period 2 will be completed in the CRC and will occur prior to RYGB or SG. The fixed study diet will be shipped by courier along with a stool collection kit. Each participant will eat the study diet on days one, two, and three of this study period. On the morning of day four, subjects present to the CRC in a fasting state and bring stool collections to the CRC. Each participant will collect three 45-minute urines with a blood sample at the midpoint of each collection. Study participants then consume a fixed breakfast and collect six 45-minute urines with blood samples in the post-prandial period.

Study period 3 will be completed in the CRC and will occur between 2 and 4 weeks post-RYGB or SG. The 2 to 4 week timing of this period was selected because the biological changes in anatomy and neuroendocrine signaling would have occurred by 2 weeks post-surgery and patients are typically advanced from a diet of soft foods to regular foods by 2 weeks. Subjects will not participate in period 3 until after clinical clearance by the surgeon for diet advancement. It is also expected that by this time any effect of anesthesia or peri-operative antibiotics and medications is minimal. The protocol of study period 3 is identical to that of period 2 with three days of study diet and CRC on day four with fasting and fed blood and urine collections (see period 2 for specifics).

Study period 4 will occur at home between 9 and 12 months post-RYGB or SG in the participant's home. The timing of this period is selected because patients have typically undergone the majority of weight loss and had time to adopt new self-chosen home diets. Urine changes expected to occur in kidney stone formers are also expected to be detectable at this time. Participants will provide a three-day diet record and complete a 1.5-hour phone call with the CRC dietician and one 24-hour urine collection (on day three). Urine collection kits will be couriered directly to home and couriered back to the Kidney Stone Lab after completion.

Study period 5 will occur in the CRC at 12 months (+/- 1 month) post-RYGB or SG. The timing of this period is selected because patients have typically undergone the majority of their weight loss and most have had resolution of metabolic syndrome. The protocol of study period 3 is identical to that of periods 2 and 3 (see period 2 for specifics).

Study Diet: Subjects will eat a diet containing 65 mmol sodium, 1740-2940mg potassium, 800-1200 mg calcium, and meals will be isocaloric with controlled macronutrient distribution. Food will be prepared in the CRC kitchen and shipped to patients. Intake of water is ad lib, other fluids only as prescribed. The diet will be prepared in consultation with dieticians, including dieticians with expertise in bariatric surgery. Food will be shipped to participants on day 1. Participants will continue to take prescribed medications and vitamin supplements per the bariatric surgery clinic.

Home diet record and nutritional data collection (study period 1, 4): Each participant will be provided a food log and a handout on portion estimates prior to home diet record. A three-day diet record will be recorded by the participant. Within one to three days of completing the diet record each participant will have a 1.5-hour phone call with the CRC dietician. The dietician will review the record for completeness and clarification, and then enter the data into the Nutritional Data System for Research (NDSR). The NDSR is a well-established, computer based, dietary analysis software program that was developed at the University of Minnesota and provides quantitative data on both micro- and macronutrients from the dietary recall. The food database in the NDSR includes over 18,000 foods and uses the United States Department of Agriculture laboratory as their primary source for nutrient values and composition. The UCM CRC has an existing contract with NDSR to support use of this software for this study.

Urine and Serum Measurements: Two 24-hour urine collections will be performed at home (with instructions provided). 24-hour urine volume, Ca, oxalate, citrate, uric acid, Na, K, Cl, Mg, sulfate, ammonium, and creatinine will be measured. Urine measurements will be performed at the University of Chicago Kidney Stone Research Group laboratory. Serum 25-vitamin D and parathyroid hormone levels will be measured through the CRC in the University of Chicago laboratory. Serum sodium, potassium, chloride, bicarbonate, calcium, phosphorus, magnesium, creatinine, and glucagon-like peptide 1 (GLP-1) will be done at the University of Chicago Kidney Stone laboratory. Serum peptide YY and insulin will be assayed at the University of Chicago Diabetes Research and Training Center laboratory. Serum glucagon will be assayed at LabCorp. Glucose will be measured using the gold standard YSI methodology at the CRC. Serum and urine will be frozen at -80 degrees C and stored at the Kidney Stone laboratory for potential later assays.

Aim 1, Urine Statistical Analysis: Urine CaOx SS will be calculated using EQUIL2 (a computer program used for the calculation of urinary saturation). We will compare the CaOx SS of men vs. women using a t-test that accounts for any differences in variances between the two groups. We will perform linear regression models by sex to determine predictors of CaOx SS. We will use Spearman's correlation tests to find independent correlations between microbial species and/or metabolic pathways with CaOx SS. Generalized linear models will be generated for any modules that are associated with high CaOx SS.

Aim 2, Stool Microbial Species and Statistical Analysis: Shotgun sequencing will be performed for all stool samples. Shotgun sequencing will be performed for all stool samples. TruSeq DNA Sample prep kit (Illumina) and reagents from KAPA Library Preparation kit (Kapa biosystems) will be used to generate libraries. Libraries will be sequenced on Illumina MiSeq platform using 2x250 nucleotide paired-end sequencing. Sequencing reads will be converted into relative abundances of microbial metabolic modules using HUMAnN and mapped to KEGG Relative abundances will be calculated using the Metagenomic Phylogenetic Analysis (MetaPhlAn) pipeline.

ELIGIBILITY:
Inclusion Criteria:

* Participants without history of stone disease, family history of stone disease
* Participants pre-bariatric surgery who are approved and planned for surgery in the Bariatric Surgery Center at University of Chicago Medicine.

Exclusion Criteria:

* Patients with primary renal diseases or renal impairment (eGFR < 90)
* Patients with known bladder voiding problems
* Patients with 25-vitamine D deficiency, as defined by level < 25ng/mL

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in urine calcium oxalate supersaturation over time | Multiple times over approximately 13 months
  Calculated using EQUIL2 from the measured urine calcium, citrate, oxalate, and volume that are directly measured in the urine

SECONDARY OUTCOMES:
Urine citrate | Multiple times over approximately 13 months (a. at the start [approximately 1 month prior to surgery] b. about 2 months in [approximately 1 month after surgery] and c. at the end [approximately 13 months from start])
  Measured directly in the urine
Calcium | Multiple times over approximately 13 months (a. at the start [approximately 1 month prior to surgery] b. about 2 months in [approximately 1 month after surgery] and c. at the end [approximately 13 months from start])
  Measured directly in the urine
Oxalate | Multiple times over approximately 13 months (a. at the start [approximately 1 month prior to surgery] b. about 2 months in [approximately 1 month after surgery] and c. at the end [approximately 13 months from start])
  Measured directly in the urine
Volume | Multiple times over approximately 13 months (a. at the start [approximately 1 month prior to surgery] b. about 2 months in [approximately 1 month after surgery] and c. at the end [approximately 13 months from start])
  Measured directly in the urine

OTHER OUTCOMES:
Association of first and secondary outcomes measures with serum insulin (physiologic parameter) | 1 day (Drawn once)
  Measured directly in the urine and blood
Association of first and secondary outcomes measures with GLP-1 (physiologic parameter) | 1 day (Drawn once)
  Measured directly in the urine and blood
Association of first and secondary outcomes measures with glucagon (physiologic parameter) | 1 day (Drawn once)
  Measured directly in the urine and blood

CONTACTS AND LOCATIONS:
Overall Officials: Prochaska Megan, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States